CLINICAL TRIAL: NCT06206226
Title: The Oh Happy Day Class - Digital Connections (OHDC-DC): an Exploratory Pilot Study
Brief Title: The Oh Happy Day Class - Digital Connections (OHDC-DC): A Pilot Study
Acronym: OHDC-DC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1437; A532007 (Other: UW- Madison); SMPH/FAMILY MED/RES GRANTS (Other: UW- Madison); Protocol Version 11/16/23 (Other: UW- Madison)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Depression; Depressive Disorder; Depressive Symptoms
Keywords: African American
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oh Happy Day Class-Digital Connections (OHDC-DC) (Experimental)
  Interventions: Behavioral: OHDC-DC

INTERVENTIONS:
Behavioral: OHDC-DC — 90-minute-weekly cognitive behavioral psycho-education classes using a mobile phone app over a 6-week period

SUMMARY:
The goal of this clinical trial is to see if a mobile phone app can deliver depression treatment to African Americans who are depressed. The main question it aims to answer is if this treatment is effective in reducing symptoms of depression.

Participants will attend six 90-minute weekly classes via an app on their phone, and will be asked to complete surveys every week. Participants can expect to be in the study for four months.

DETAILED DESCRIPTION:
The Oh Happy Day Class-Digital Connections (OHDC-DC) is designed for African American adults experiencing clinical depression (CD). OHDC originally comprised of 13 treatment modules focused on culturally relevant strategies to increase knowledge of depression and healthy coping behaviors aimed at reducing symptoms of clinical depression and improving health outcomes.

The Oh Happy Day Class-Digital Connections (OHDC-DC) comprise of 5 core elements of the OHDC-DC:

1. 90-minute-weekly cognitive behavioral psycho-education classes over a 6-week period.
2. Six classes will be offered and facilitated online in the computerized OHDC-DC.
3. Participants will be encouraged to stay engaged between classes by digitally connecting on the app with the class content. On the app they will receive reminders and messages from staff and participants to stay digitally connected and engaged.
4. Embedded in the classes and content is psychoeducation with an emphasis on educating participants about depression, raising awareness of mental illness with the goal of normalizing it and reducing stigma, and increasing healthy coping behaviors, and.
5. The intervention will be delivered by a licensed mental health clinician.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* Age 18 and older
* Experiencing depression (as evidenced by a score of 5 or higher on the PHQ-9)
* Own a mobile phone

Exclusion Criteria:

* Individuals who are currently receiving psychotherapy
* Individuals who are presently experiencing suicidal ideation
* Individuals who started psychotropic medication less than three months prior to the start of the OHDC will be excluded from the study
* Participants scoring 25 or higher on the PHQ-9 will be screened out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Personal Health Questionnaire Depression Scale score | Baseline to one month post-intervention (approximately 12 weeks)
  Using the 8 item Personal Health Questionnaire Depression Scale (PHQ-8), participants will rate how much they have been bothered by symptoms on a scale of 0-3 with a possible range of 0 to 24. Higher scores indicate greater degree of depression.
Change in Generalized Anxiety Disorder 7-item (GAD-7) score | Baseline to one month post-intervention (approximately 12 weeks)
  Using the GAD-7 score, participants will rate how much they have been bothered by symptoms on a scale of 0-3 with a possible range of 0 to 24. Higher scores indicate greater degree of anxiety.
Change in Quick Inventory of Depressive Symptomatology (QIDS) | Baseline to one month post-intervention (approximately 12 weeks)
  Using the 16-item QIDS, participants will rate how much they have been bothered by symptoms on a scale of 0-3 with a possible range of 0 to 27. Higher scores indicate greater degree of depression.
Satisfaction with intervention | 12 weeks
  Participants will rate their satisfaction with the intervention by answering a 9-item questionnaire with a scale of 1-7 (1= none of the time, 7= all of the time). Higher scores indicate greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Earlise Ward, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No